CLINICAL TRIAL: NCT07332195
Title: Clinical and Radiographic Analysis of Implant Rehabilitations in a Hospital Setting: a Prospective Study
Brief Title: Implant Rehabilitations in a Hospital Setting
Status: Not yet recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: ID 7698
Record Dates: First submitted 2025-11-18; First posted 2026-01-12 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2025-11

CONDITIONS: Patients Requiring an Implant-supported Rehabilitation; Edentulous Patients Requiring an Implant-supported Rehabilitation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Implant-supported rehabilitation: Patients aged >18 years who require implant-supported rehabilitation

SUMMARY:
Dental implants are considered a predictable rehabilitation option for tooth extraction or missing teeth. The use of dental implants has evolved into a viable prosthetic alternative to conventional tooth-supported fixed prostheses or removable dentures, with advantages in terms of patient satisfaction and quality of life. Long-term studies have reported excellent success and survival rates for implants used in prosthetic rehabilitation. Benefits in terms of patient satisfaction and preservation of adjacent tooth structure are among the advantages of implant-supported restorations over prosthetic alternatives. However, dental implants can be subject to mechanical and biological complications. After the first year of function, marginal bone loss is minimal around most oral implants. Nevertheless, marginal bone loss or the onset of bacterial-related biological complications, such as mucositis and peri-implantitis, can occur. Despite the growing number of publications in the field of implant rehabilitation, to date only a few studies have investigated the outcomes of implant rehabilitation in a hospital setting characterized by patients with concomitant or previous systemic therapies and pathologies. The objective of this study is to evaluate the success of implant therapy, peri-implant marginal bone resorption (MBL), clinical parameters of peri-implant health, aesthetic parameters of rehabilitation, and patient-reported treatment outcomes in a sample of patients treated in a hospital setting.

ELIGIBILITY:
Inclusion Criteria:

* Patients requiring implant surgery for edentulous rehabilitation;
* Age > 18;
* Achievement of FMPS and FMBS ≤ 15%;
* Signed written informed consent to participate in the study.

Exclusion Criteria:

* Uncontrolled diabetes or hypertension;
* Uncontrolled periodontal disease;
* Inability to perform consistent and continuous follow-up;
* Pregnancy or breastfeeding;
* Inability to provide written informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged >18 years who require implant-supported rehabilitation
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2030-12-01 (Estimated); Study Completion 2030-12-01 (Estimated)

PRIMARY OUTCOMES:
Peri-implant marginal bone loss | From Implant placement to 5 year follow up.
  Measurements were performed in millimeters using intraoral radiographs.
Implant survival rate | From Implant placement to 5 year follow up.
  Rate of dental implants remaining in situ, measured as a proportion.

SECONDARY OUTCOMES:
Implant success rate | From Implant placement to 5 year follow up.
  Absence of biological and technical complications, expressed as a proportion.
Prosthesis survival rate | From Implant placement to 5 year follow up.
  Rate of prostheses remaining in situ, expressed as a proportion.
Prosthesis success rate | From Implant placement to 5 year follow up.
  Absence of technical complications, expressed as a proportion.
Esthetic evaluation | From Implant placement to 5 year follow up.
  Assessed using the PES/WES esthetic index. Scores range from 0 to 14 for the PES and from 0 to 10 for the WES, with higher scores indicating better esthetic outcomes.
Patient-Reported Outcome Measures | From Implant placement to 5 year follow up.
  Recorded using a specifically designed questionnaire and measured with a visual analogue scale (VAS) ranging from 0 to 10, with higher scores indicating better outcomes.
Volumetric analysis | From Implant placement to 5 year follow up.
  Assessed by superimposing the baseline volume with the volume recorded during follow-up using intraoral scans, measured in cubic millimeters.
Glycated hemoglobin level | From Implant placement to 5 year follow up.
  Analysis of glycated hemoglobin levels recorded at baseline and during follow-up.
Diabetes | From Implant placement to 5 year follow up.
  Analysis of the influence of diabetes during follow-up.
Influence of medications relevant to bone/tissue metabolism | From Implant placement to 5 year follow up.
  Analysis of the influence of medications relevant to bone and tissue metabolism.
Osteoporosis | From Implant placement to 5 year follow up.
  Analysis of influence of osteoporosis.
Cardiovascular disease | From Implant placement to 5 year follow up.
  Analysis of influence of cardiovascuar disease.
Complete Blood Count | From Implant placement to 5 year follow up.
  Analysis of the influence of complete blood count parameters.

CONTACTS AND LOCATIONS:
Overall Officials: Carlo Lajolo, Principal Investigator — Fondazione Policlinico Universitario A. Gemelli, IRCCS

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chen ST, Buser D. Clinical and esthetic outcomes of implants placed in postextraction sites. Int J Oral Maxillofac Implants. 2009;24 Suppl:186-217. PMID 19885446
- [Background] Gelb DA. Immediate implant surgery: three-year retrospective evaluation of 50 consecutive cases. Int J Oral Maxillofac Implants. 1993;8(4):388-99. PMID 8270307
- [Background] Nir-Hadar O, Palmer M, Soskolne WA. Delayed immediate implants: alveolar bone changes during the healing period. Clin Oral Implants Res. 1998 Feb;9(1):26-33. doi: 10.1034/j.1600-0501.1998.090104.x. PMID 9590942
- [Background] Adell R, Lekholm U, Rockler B, Branemark PI. A 15-year study of osseointegrated implants in the treatment of the edentulous jaw. Int J Oral Surg. 1981 Dec;10(6):387-416. doi: 10.1016/s0300-9785(81)80077-4. PMID 6809663
- [Background] 3) Branemark PI. Introduction to osseointegration. In: BranemarkPI, Zarb GA, Albrektsson T, Rosen HM, eds. Tissue-IntegratedProstheses: Osseointegration in Clinical Dentistry. Chicago:Quintessence Publishing Company, Inc; 1985:11-76.
- [Background] den Hartog L, Slater JJ, Vissink A, Meijer HJ, Raghoebar GM. Treatment outcome of immediate, early and conventional single-tooth implants in the aesthetic zone: a systematic review to survival, bone level, soft-tissue, aesthetics and patient satisfaction. J Clin Periodontol. 2008 Dec;35(12):1073-86. doi: 10.1111/j.1600-051X.2008.01330.x. PMID 19040585
- [Background] Siadat H, Alikhasi M, Beyabanaki E. Interim Prosthesis Options for Dental Implants. J Prosthodont. 2017 Jun;26(4):331-338. doi: 10.1111/jopr.12421. Epub 2016 Jan 24. PMID 26805651